CLINICAL TRIAL: NCT06154044
Title: The Effects of Cell Therapy on Myocardial Recovery in Chronic Heart Failure Patients Undergoing Left Ventricular Assist Device Support: A Pilot Trial (CELL-VAD Pilot)
Brief Title: Cell Therapy and Myocardial Recovery in Heart Failure Patients Undergoing Left Ventricular Assist Device Support
Acronym: CELL-VAD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMC 1
Record Dates: First submitted 2023-11-06; First posted 2023-12-01 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Mechanical Circulatory Support
Keywords: heart failure; mechanical circulatory support; stem cells
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Masking Description: Imaging core lab employees will be blinded to the patient's status (before or after cell therapy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): After successful LVAD implantation, patients will be enrolled and followed for 2 months to allow for postoperative rehabilitation and heart failure medical therapy and LVAD support optimization. All patients will then undergo autologous CD34+ cell therapy which will be delivered via intracoronary route. All patients will be followed for 6 months after cell therapy. At baseline, and at 1, 3 and 6 months after cell therapy, we will perform comprehensive clinical evaluation. Clinical, biochemical, biomarker-related, imaging and myocardial histology data will be transferred to a secured central database.
  Interventions: Biological: CD34+ stem cell therapy

INTERVENTIONS:
Biological: CD34+ stem cell therapy — After 5-days GCSF stimulation all patients will undergo apheresis to obtain CD34+ cell which will subsequently be injected in the target coronary artery using microcatheter.

SUMMARY:
The goal of CELL-VAD Pilot trial is to investigate a personalized stem cell therapy approach for patients with advanced non-ischemic chronic heart failure (NICM) who are supported by LVAD. In the clinical trial, the investigators aim to enroll 10 patients with NICM, scheduled for LVAD implantation. After successful LVAD implantation, patients will be enrolled and followed for 2 months to allow for postoperative rehabilitation and heart failure medical therapy and LVAD support optimization. All patients will then undergo autologous CD34+ cell therapy which will be intracoronaryly delivered to the target myocardium using NOGA electromechanical mapping system. All patients will be followed for 6 months after cell therapy. At baseline, and at 1, 3, and 6 months after cell therapy, the investigators will perform comprehensive clinical evaluation.

DETAILED DESCRIPTION:
PROBLEM IDENTIFICATION Left ventricular assist device (LVAD) technology has evolved significantly and represents a standard of care for patients with advanced chronic heart failure. However, a significant discrepancy exists between structural and functional recovery of the failing myocardium, as only a small fraction (2%) of LVAD-supported patients demonstrate reverse structural remodeling and eventually reach clinically significant and stable functional improvement that allows for LVAD removal. Thus, there is a significant unmet need to define better the mechanisms of myocardial reverse remodeling in advanced chronic heart failure patients undergoing LVAD support.

OBJECTIVES

The goal of CELL-VAD Pilot trial is to investigate a personalized stem cell therapy approach for patients with advanced non-ischemic chronic heart failure (NICM) who are supported by LVAD. The investigators propose a Phase II non-randomized single-center clinical study focusing on (1) the administration of stem cell therapy that would allow for durable improvements in heart function and structure in NICM-LVAD patients. By using integrated analysis of multimodality imaging and biomarkers of fibrosis and angiogenesis, this project aims to (2) better define the pathophysiological mechanisms involved in myocardial recovery. Additionally, the investigators also aim to (3) define the safety parameters of stem cell therapy in NICM-LVAD patients. Based on these aims, the specific objectives of the CELL-VAD Pilot trial are:

The primary objective of this study is to investigate the safety and efficacy of stem cell therapy in NICM-LVAD patients, by evaluating changes in left ventricular structure and function, biomarkers of neurohormonal activation, patient exercise capacity, and clinical outcome.

The secondary objective of this study is to better define pathophysiological mechanisms involved in myocardial recovery in NICM-LVAD patients, by evaluating temporal changes in myocardial perfusion and in biomarkers of myocardial fibrosis in angiogenesis.

STUDY DESIGN The CELL-VAD Pilot trial consists of a clinical trial (WP1) and a multimodality imaging platform (WP2). The overall duration of the project is 3 years (36 months).

In the clinical trial, the investigators aim to enroll 10 patients with NICM, scheduled for LVAD implantation. After successful LVAD implantation, patients will be enrolled and followed for 2 months to allow for postoperative rehabilitation and heart failure medical therapy and LVAD support optimization. All patients will then undergo autologous CD34+ cell therapy which will be delivered via the intracoronary route. All patients will be followed for 6 months after cell therapy. At baseline, and at 1, 3, and 6 months after cell therapy, the investigators will perform comprehensive clinical evaluation. Clinical, biochemical, biomarker-related, imaging, and myocardial histology data will be transferred to a secured central database.

The investigators also aim to develop a personalized multimodality imaging platform by integrating the data obtained from advanced echocardiography and PET imaging.

EXPECTED OUTCOMES The investigators expect to demonstrate that in NICM-LVAD patients transendocardial autologous CD34+ cell therapy is safe and efficient, promoting the structural and functional reverse remodelling of the failing myocardium. Additionally, the results of this trial will establish a solid framework of knowledge and expertise for future clinical trials to build on.

ELIGIBILITY:
Patient inclusion criteria will consist of all of the following:

1. non-ischemic dilated cardiomyopathy
2. patient accepted for LVAD support
3. optimal (or maximal tolerable therapy) heart failure ≥ 2 months
4. age 18-65 years
5. ability to provide informed consent

Patient exclusion criteria will consist of any of the following:

1. ischemic cardiomyopathy
2. Cardiomyopathy with a reversible cause that has not been treated e.g. thyroid disease, alcohol abuse, hypophosphataemia, hypocalcaemia, cocaine abuse, selenium toxicity & chronic uncontrolled tachycardia.
3. Cardiomyopathy in association with a neuromuscular disorder e.g. Duchenne's progressive muscular dystrophy.
4. ongoing or recent (less than 1 month) infection
5. acute multi-organ failure
6. clinically significant anemia (Hb < 10 g/dL)
7. clinically significant leukopenia (L < 2 x 109/L) or leukocytosis (L > 14 x 109/L)
8. clinically significant thrombocytopenia (TRC < 50 x 109/L)
9. known disorders of hemostasis that can not be corrected
10. history of any thromboembolic complications
11. chronic kidney disease (higher than stage III)
12. chronic liver disease (Child B or C)
13. diminished functional capacity for other reasons such as COPD, moderate or severe claudications, severe musculosceletal system pain or morbid obesity (BMI > 35 kg/m2)
14. aortic stenosis (AVA < 1.3 cm2) or ocluded aortic valve
15. artificial (mechanical or biological) aortic valve
16. patients with reduced immune response
17. history of limphoprolipherative disorders or malignancy within 5 years
18. left ventricular thrombus
19. participation in another interventional clinical trial
20. life expectancy less than 12 months
21. known hypersensitivity to DMSO, penicillin or streptomycin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
change in left ventricular ejection fraction (LVEF) | Baseline to 6 months
  change in left ventricular ejection fraction (LVEF), measured by transthoracic echocardiography using Simpson's rule between the time of stem cell therapy and 6 months.
Changes in left ventricular end-systolic and end-diastolic dimensions | Baseline to 3 and 6 months
  Changes in left ventricular end-systolic (LVESd) and end-diastolic dimensions (LVEDd) measured by transthoracic echocardiography in parasternal longitudinal axis with expected change > 10%.
Changes in left ventricular longitudinal and circumferential strains | Baseline to 3 and 6 months
  Changes in left ventricular longitudinal and circumferential strains will be measured using transthoracic echocardiography and segmental wall motion analysis with expected change > 10%.
Changes in right ventricular size | Baseline to 3 and 6 months
  Changes in right ventricular size (RVIDd) will be measured using transthoracic echocardiography with expected change > 10%.
Change in serum neurohumoral activation | Baseline to 3 and 6 months
  Change in serum neurohumoral activation will be assessed measuring NT-proBNP serum levels, with expected decrease > 30%.
Changes in serum markers of fibrosis and angiogenesis | Baseline to 3 and 6 months
  Changes in serum markers of fibrosis and angiogenesis will be assessed by measuring biomarkers of fibrosis and angiogenesis using Luminex commercially available kits (Human XL Cytokine Luminex® Performance Assay 46-plex); any detectable change will be considered a positive response.
Change in 6-minute walk test | Baseline to 3 and 6 months
  Change in 6-minute walk test with expected increase > 30 m
Change in quality of life questionnaire score | Baseline to 3 and 6 months
  Change in quality of life KCCQ questionnaire score with expected decrease of ≥ 5 points
Change in heart failure-related hospitalization | Baseline to 3 and 6 months
  Change in heart failure-related hospitalization; any decrease will be considered

CONTACTS AND LOCATIONS:
Overall Officials: Bojan Vrtovec, MD, PhD, Principal Investigator — UMC Ljubljana
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided